CLINICAL TRIAL: NCT02446067
Title: Cerebral Hemodynamics With rTMS in Alcohol Dependence: A Randomized, Sham Controlled Study
Brief Title: Cerebral Hemodynamics With rTMS in Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Psychiatry, Ranchi, India (Other)
Responsible Party: Principal Investigator, Dr. Biswa Ranjan Mishra, Senior resident, Central Institute of Psychiatry, Ranchi, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPRanchi
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Alcohol Dependence
Keywords: Transcranial Doppler (TCD) sonography; rTMS; Cerebral hemodynamics
MeSH Terms: conditions — Alcoholism; Choroideremia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy control (No Intervention): No Repetitive Transcranial Magnetic Stimulation (rTMS)
- Active rTMS group (Active Comparator): Active Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham rTMS group (Sham Comparator): Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — The motor threshold for the left abductor pollicis brevis was determined using a figure-of-eight-shaped coil at 1 Hz frequency. Ten (over 2 weeks) rTMS sessions were administered over the right dorsolateral prefrontal cortex with an air-cooled figure-of-eight coil, angled tangentially to the head. At right DLPFC, active high-frequency (10 Hz) stimulation was administered for 4.9 seconds per train, with inter-train interval of 30 seconds, and a total of 20 trains per session. Each patient received 1000 pulses per day. The sham group was administered rTMS with the same parameters, but using a figure-of-eight sham coil.
  Arms: Active rTMS group; Sham rTMS group

SUMMARY:
The present study measures the cerebral hemodynamic indices of alcohol dependent patients and observe the relative changes in these parameters with rTMS application.

DETAILED DESCRIPTION:
Alcohol abuse is a worldwide problem causing serious physical, psychological, social and economic consequences. Chronic alcohol intake has been found to increased blood viscosity, erythrocyte deformability or dehydration resulting in alterations of cerebral blood flow measures. Transcranial Doppler (TCD) sonography is a non-invasive radiological tool used for assessing the hemodynamics of the basal cerebral arteries, which can thus indirectly reflect the relative changes in regional cerebral blood flow velocity (CBFV) and vascular wall resistance. It has been used to evaluate the relative cerebral blood flow velocity changes in various psychiatric disorders like depression, schizophrenia, panic disorder, and substance use disorders including alcohol and marijuana. TCD also gives a real time assessment of the abrupt or short and long lasting effects of any external mechanical manipulation or functional stimulation of the intracranial circulation.

The Mean flow velocity (MV) is the average of the edge frequency over a cardiac cycle; the edge frequency being the envelope of instantaneous peak velocities throughout the course of a cardiac cycle. Pulsatility index (PI) represents an estimate of downstream vascular resistance; low resistance vascular beds have higher diastolic flow velocities than high resistance vascular beds, hence they have low PI, and vice versa. Similarly, Resistance index (RI) is another presumptive measure of downstream vascular resistance.

TCD sonography studies in alcoholism have revealed reduced mean blood flow velocities in basal cerebral arteries in chronic alcohol dependence, [1] as well as in acute stage of intoxication, but an increase after resolution of withdrawal state. [12] However, ethanol in low concentration has been found to increase the systolic, diastolic and mean blood flow velocity in middle cerebral arteries (MCA), anterior cerebral arteries (ACA) and decrease the resistance indices by reducing the cerebrovascular resistance in healthy individuals. Studies have reported that alcohol related hepatic dysfunction results in increased blood viscosity and reduced velocity in the cerebral arteries, which can be a risk factor for ischemic brain diseases. So, normalization of hemodynamic parameters is important in the prevention of possible ischemic brain diseases due to alcohol dependence.

Studies evaluating cerebral hemodynamic response to rTMS application have been limited to healthy individuals, with high frequency rTMS application found to increase the cerebral blood flow velocities in both anterior and posterior basal cerebral arteries, and low frequency rTMS to temporarily decrease the blood flow velocity in ipsilateral MCA followed by an increase in the contralateral MCA. With this background, the present study was conducted to measure the cerebral hemodynamic indices of alcohol dependent patients and observe the relative changes in these parameters with rTMS application.

ELIGIBILITY:
Inclusion Criteria:

* Right handed, male patients, aged between 18-60 years, with diagnosis of alcohol dependence according to DSM-IV TR, after resolution of withdrawal symptoms i.e. having Clinical Institute of Withdrawal Assessment in Alcohol Withdrawal (CIWA-Ar) score of ≤10, were included in the study.

Exclusion Criteria:

* Patients with comorbid psychiatric, major medical or neurological disorders or with a pacemaker or metal in any part of the body were excluded from the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Mean velocity (MV) of middle cerebral artery (MCA) and anterior cerebral artery (ACA) | up to 5 minutes after last (10th) rTMS session

SECONDARY OUTCOMES:
Pulsatility index (PI) of middle cerebral artery (MCA) and anterior cerebral artery (ACA) | up to 5 minutes after last (10th) rTMS session
Resistance index (RI) of middle cerebral artery (MCA) and anterior cerebral artery (ACA) | up to 5 minutes after last (10th) rTMS session

CONTACTS AND LOCATIONS:
Locations (1):
- Central Institute of Psychiatry, Ranchi, Jharkhand, India

REFERENCES:
- [Result] Gdovinova Z. Blood flow velocity in the middle cerebral artery in heavy alcohol drinkers. Alcohol Alcohol. 2001 Jul-Aug;36(4):346-8. doi: 10.1093/alcalc/36.4.346. PMID 11468137
- [Result] Pecuch PW, Evers S, Folkerts HW, Michael N, Arolt V. The cerebral hemodynamics of repetitive transcranial magnetic stimulation. Eur Arch Psychiatry Clin Neurosci. 2000;250(6):320-4. doi: 10.1007/s004060070007. PMID 11153967
- [Result] de Castro AG, Bajbouj M, Schlattmann P, Lemke H, Heuser I, Neu P. Cerebrovascular reactivity in depressed patients without vascular risk factors. J Psychiatr Res. 2008 Jan;42(1):78-82. doi: 10.1016/j.jpsychires.2006.10.001. Epub 2006 Nov 20. PMID 17113598
- [Result] Mathew RJ, Wilson WH. Substance abuse and cerebral blood flow. Am J Psychiatry. 1991 Mar;148(3):292-305. doi: 10.1176/ajp.148.3.292. PMID 1992832
- [Result] Gdovinova Z. Cerebral blood flow velocity and erythrocyte deformability in heavy alcohol drinkers at the acute stage and two weeks after withdrawal. Drug Alcohol Depend. 2006 Feb 28;81(3):207-13. doi: 10.1016/j.drugalcdep.2005.07.006. Epub 2005 Aug 29. PMID 16129568
- [Result] Blaha M, Aaslid R, Douville CM, Correra R, Newell DW. Cerebral blood flow and dynamic cerebral autoregulation during ethanol intoxication and hypercapnia. J Clin Neurosci. 2003 Mar;10(2):195-8. doi: 10.1016/s0967-5868(02)00126-1. PMID 12637048
- [Result] Stendel R, Irnich B, al Hassan AA, Heidenreich J, Pietilae T. The influence of ethanol on blood flow velocity in major cerebral vessels. A prospective and controlled study. Alcohol. 2006 Apr;38(3):139-46. doi: 10.1016/j.alcohol.2006.06.005. Epub 2006 Jul 28. PMID 16905439
- [Result] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811